CLINICAL TRIAL: NCT05875753
Title: Preliminary Study of 68Ga-FAPI-FS PET/CT in Patients With Pancreatic Cancer
Brief Title: 68Ga-FAPI-FS PET/CT and PET/MR in Pancreatic Cancer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FAPI-FS
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Pancreatic Cancer
Keywords: 68Ga-FAPI-FS; PET/CT
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-FAPI-FS PET/CT (Experimental): Each patient will receive one dose of 68Ga-FAPI-FS by intravenous route. Dedicated whole-body PET/CT imaging will be performed.
  Interventions: Diagnostic Test: 68Ga-FAPI-FS PET/CT

INTERVENTIONS:
Diagnostic Test: 68Ga-FAPI-FS PET/CT — Participants will be administered a single, intravenous bolus of 68Ga-FAPI-FS. The recommended administered activity of 68Ga-NY104 is 1.8-2.2 MBq per kilogram bodyweight, subject to variation that may be required owing to variable elution efficiencies obtained during the lifetime of the 68Ga / 68Ga generator.
  The CT and PET imaging session will begin approximately 45 to 75 minutes after 68Ga-FAPI-FS administration.

SUMMARY:
This is a preliminary study of 68Ga-FAPI-FS PET/CT or PET/MR in patients with confirmed or suspicious pancreatic cancer. The goal is to determine the safety, biodistribution, and tumor uptake of 68Ga-FAPI-FS.

DETAILED DESCRIPTION:
This is a preliminary phase 0 study in patients with confirmed or suspicious pancreatic cancer. Each patient will receive one dose of 68Ga-FAPI-FS by intravenous route. Dedicated whole-body PET/CT imaging will be performed. A comparative 18F-FDG PET/CT will also be performed within a week.

ELIGIBILITY:
Inclusion Criteria:

1. Pancreatic cancer confirmed by histopathological results or pancreatic lesions with typical radiological appearance.
2. Expected survival of at least 3 months
3. ECOG ≤ 2
4. Written informed consent provided for participation in the trial
5. In the opinion of investigator, willing and able to comply with required study procedures.

Exclusion Criteria:

1. Pregnancy or breastfeeding.
2. Severe claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events after injection of 68Ga-FAPI-FS | From tracer injection to 3 hour post-injection
  Adverse events will be recorded according to CTCEA v4.03

SECONDARY OUTCOMES:
SUVmax of liver on 68Ga-FAPI-FS | From study completion to 1 month after completion
  The liver uptake will be measured using SUVmax with a 40% threshold.
SUVmax of normal pancreas on 68Ga-FAPI-FS | From study completion to 1 month after completion
  The normal pancreas uptake will be measured using SUVmax with a 40% threshold.
SUVmax of blood pool on 68Ga-FAPI-FS | From study completion to 1 month after completion
  The blood pool uptake will be measured using SUVmax with a 40% threshold.
SUVmax of lung on 68Ga-FAPI-FS | From study completion to 1 month after completion
  The lung uptake will be measured using SUVmax with a 40% threshold.
SUVmax of brain on 68Ga-FAPI-FS | From study completion to 1 month after completion
  The brain uptake will be measured using SUVmax with a 40% threshold.
SUVmax of muscle on 68Ga-FAPI-FS | From study completion to 1 month after completion
  The muscle will be measured using SUVmax with a 40% threshold.
SUVmax of tumor lesions on 68Ga-FAPI-FS | From study completion to 1 month after completion
  The tumor lesions will be measured using SUVmax with a 40% threshold.

CONTACTS AND LOCATIONS:
Overall Officials: Li Huo, MD, Principal Investigator — Peking Uion Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No